CLINICAL TRIAL: NCT01861366
Title: Clinical Outcome in Nursing Home Residents After Implementation of Nutritional Guidelines
Brief Title: Implementation of Nutritional Guidelines and Effects in Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MuMs07
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Implementation Strategies; Nutritional Outcome of Nursing Home Residents
Keywords: Implementation; Guidelines; Nutrition; Nursing home

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- External facilitator (Experimental): The external facilitation is a one year multifaceted intervention, including support, guidance, practice audit and feedback, training targeted to a team of practitioners involving the unit manager, the nurses and diet aides at the nursing home. The facilitator is a researcher and dietician.
  Interventions: Other: A one year multifaceted implementation strategy
- Educational outreach visit (Active Comparator): The outreach visit is a three hour lecture about the nutritional guidelines targeted to a team of practitioners including the unit manager, the nurses and diet aides at the nursing home. The trained person giving the lecture is a researcher and dietician.
  Interventions: Other: A three hour lecture about the guidelines

INTERVENTIONS:
Other: A one year multifaceted implementation strategy
  Arms: External facilitator
Other: A three hour lecture about the guidelines
  Arms: Educational outreach visit

SUMMARY:
The aim of this study is to examine two implementation strategies (external facilitation and educational outreach visit) when introducing nutritional guidelines in the elderly care setting and to evaluate the results of the implementation by clinical outcome measures of the nursing home residents.

The hypothesis is that the residents affected by the external facilitation strategy will stay stable in the measured clinical outcomes, while the residents influenced by the educational outreach visit will deteriorate during the implementation process.

ELIGIBILITY:
Inclusion Criteria:

* age of 65 or older
* nursing home resident
* persons who manage the examination methods (interviews and blood samples)

Exclusion Criteria:

- persons in terminal stage of life

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Nutritional status | 2 years
  Nutritional status is assessed with the Mini Nutritional Assessment-Short Form tool

SECONDARY OUTCOMES:
Functional status | 2 years
  Functional status is assessed with ADL (Activities in Daily Living) Barthel index.
Cognitive status | 2 years
  Cognitive status is assessed with Short Portable Mental Status Questionnaire (SPMSQ).
Health-related Quality of Life | 2 years
  Health-related Quality of Life is assessed with EQ-5D.

OTHER OUTCOMES:
Biochemical markers | 2 years
  Blood samples are collected for analysis of vitamin D, albumin, CRP (C-reactive protein), insulin-like growth factor 1 (IGF-1), creatinine and cystatin C, which gives biochemical information on the nutritional status, inflammation activity and renal function.
Morbidity | 2 years
  Morbidity is assessed with Charlson Comorbidity Index (CCI).

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Cederholm, Prof, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Derived] Torma J, Winblad U, Saletti A, Cederholm T. Strategies to implement community guidelines on nutrition and their long-term clinical effects in nursing home residents. J Nutr Health Aging. 2015 Jan;19(1):70-6. doi: 10.1007/s12603-014-0522-4. PMID 25560819